CLINICAL TRIAL: NCT04660942
Title: Child Development and Genetic Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001521A3
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy child
- Experimental: Patients with developmental delay

SUMMARY:
A study of the relation between genetic biomarkers and child development in Taiwan.

DETAILED DESCRIPTION:
The interaction between gene and environment (G×E) can be a very complicated process that influences child development. As a pilot study of child development biomarkers, this study investigates genes related to child development.

ELIGIBILITY:
Inclusion Criteria of Healthy Child:

* Age 2-18 y/o
* Agree to sign informed consent

Exclusion Criteria of Healthy Child:

* Central nervous system disease
* Neuromuscular Disorders
* Congenital Abnormality
* Genetic Disease
* Dysesthesia
* Hearing Impairment

Inclusion Criteria of Child with developmental delay:

* Patients with Language Disorder
* Age 2-18 y/o
* Agree to sign informed consent

Exclusion Criteria of Child with developmental delay:

* Hearing Impairment

Inclusion Criteria of Adult:

* His or her child participated in this study, and gene abnormality was found.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy children, children with developmental delay and adults whose children had gene abnormality were recruited.
Sampling Method: Probability Sample
Enrollment: 446 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Scores of cognitive function 1 | baseline
  Bayley Scales of Infant and Toddler Development (Scores from 0 to 140, higher scores mean a better outcome.)
Scores of cognitive function (2 y/o to 6 y/o) | baseline
  Wechsler Preschool and Primary Scale of Intelligence (Scores from 0 to 200, higher scores mean a better outcome.)
Scores of cognitive function (6 y/o to 16 y/o) | baseline
  Wechsler Intelligence Scale for Children (Scores from 0 to 200, higher scores mean a better outcome.)
Scores of cognitive function 3 | baseline
  Test of Nonverbal Intelligence-Fourth Edition (Scores from 0 to 60, higher scores mean a better outcome.)
Scores of cognitive psychological function | baseline
  Cantab MOT, PAL, SWM, SOC tests
Scores of language function | baseline
  Peabody Picture Vocabulary Test-Revised (Scores from 0 to 124, higher scores mean a better outcome.)
Scores of language function 2 | baseline
  Preschool Language Impaired Scale(PLS)/Language Impaired Scale(LS) (PLS: Scores from 0 to 65, higher scores mean a better outcome. LS: Scores from 0 to 73, higher scores mean a better outcome.)
Scores of general development | baseline
  Comprehensive Developmental Inventory for Infants and Toddlers (Higher scores mean a better outcome.)
Scores of social behavior 1 | baseline
  Clancy Behavior Scale (Scores from 0 to 42, lower scores mean a better outcome.)
Scores of social behavior 2 | baseline
  Swanson, Nolan, and Pelham, Version IV (Lower scores mean a better outcome.)
Scores of motor ability 1 | baseline
  The Berry-Buktenica Developmental Test of Visual-Motor Integration (Scores from 0 to 81, Higher scores mean a better outcome.)
Scores of motor ability 2 | baseline
  Measure of Grip and Grasp (Higher scores mean a better outcome.)
Gene test (Mircoarray) | baseline
  Microarray (Use Axiom Genome-Wide TWB 2.0 Array Plate (TWB 2.0) to analyze SNPs of disease-related biomarkers.)
Gene test (WES1) | baseline
  Whole-Exome Sequencing (Use Burrows-Wheeler Aligner (BWA) 85 to screen out the variant discovery and genotyping.)
Gene test (WES2) | baseline
  Whole-Exome Sequencing (Use Samtools86 to screen out the variant discovery and genotyping.)
Gene test (WES3) | baseline
  Whole-Exome Sequencing (Use Picard to screen out the variant discovery and genotyping.)
Gene test (WES4) | baseline
  Whole-Exome Sequencing (Use Genome Analysis Toolkit (GATK) to screen out the variant discovery and genotyping.)

SECONDARY OUTCOMES:
Scores of participation(2-5 y/o) | baseline
  Assessment of Preschool Children's Participation (Scores from 0 to 45, higher scores mean a better outcome.)
Scores of participation(>6 y/o) | baseline
  Children Assessment of Participation and Enjoyment and Preferences for Activity of Children (Higher scores mean a better outcome.)
Scores of activities | baseline
  Functional Independence Measure for Children (Scores from 18 to 126, higher scores mean a better outcome.)
Scores of quality of life | baseline
  Pediatric Quality of Life Inventory TM (Scores from 0 to 102, higher scores mean a better outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, Phd, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan